**Protocol title:** Safety, feasibility and efficacy of vitamin D supplementation in women with metastatic breast cancer (SAFE-D)

**NCT:** 02186015

Date: November 14, 2018

**Protocol title:** Safety, feasibility and efficacy of vitamin D supplementation in women with metastatic breast cancer (SAFE-D)

Principal Investigator: Patricia Sheean, PhD, RD

**Research Team:** William Adams, MS; Cara Joyce, PhD, Sue Penckofer, PhD, RN; Ruta Rao, MD; Patricia Robinson, MD;

## **Statistical Analyses Conducted**

Descriptive statistics were conducted to examine differences in sociodemographics, medical characteristics and dietary intake stratified by sufficient vs. insufficient serum 25(OH)D at baseline. Statistical differences between groups were assessed with Wilcoxon rank sum tests for continuous variables and chi-square or Fisher's exact test for nominal variables. Among those treated with 8 weeks of high dose cholecalciferol, changes from baseline were assessed with Wilcoxon signed rank tests for continuous scores. Analyses were performed with SAS version 9.4 (Cary, NC). A p value of <0.05 was used to denote statistical significance and based on the exploratory nature of this study, a p value of <0.10 was used to designate statistical trends.